CLINICAL TRIAL: NCT03707860
Title: Radiation Oncology Mobile Application: Symptoms Reporting System and Quality Assurance Tool
Brief Title: Radiation Oncology Mobile Application
Acronym: γ-App
Status: Withdrawn | Type: Observational
Why Stopped: the program couldn't be implemented
Sponsor: King Hussein Cancer Center (Other)
Responsible Party: Principal Investigator, Ramiz Abu-Hijlih, Consultant Radiation Oncology, King Hussein Cancer Center
Other Study IDs: 18 KHCC 86
Record Dates: First submitted 2018-10-12; First posted 2018-10-16 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Head and Neck Cancer; Radiation Toxicity
MeSH Terms: conditions — Head and Neck Neoplasms; Radiation Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- head and neck radiotherapy patients: (Single arm); Patients receiving radiotherapy for head and neck cancers can report their symptoms through the mobile app.

SUMMARY:
To develop a novel a mobile phone application (available on Android and IOS) for patients receiving radiation treatment for head and neck cancer. Through this application, patients will get access to their treatment calender, through a system connected with Mosiac database, which provides a timely and precise access to their treatments schedule.

In addition, patients will be able to report their treatment related toxicity in real time fashion, these symptoms will be addressed daily instead of the weekly floor clinic checks.

Furthermore, the radiation oncologist will receive an instant notification through the application, if there is error in patient's treatment (missing field, wrong dose, etc..)

ELIGIBILITY:
Inclusion Criteria:

Adult patients receiving definitive or adjuvant RT to head and neck site Chemotherapy is allowed PS:0-1 Has a smart phone

Exclusion Criteria:

Poor performance early laryngeal cancer Patient with metastatic disease, or palliative intent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to our radiation oncology clinic with head and neck cancer.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-10-20 (Actual); Study Completion 2021-10-20 (Actual)

PRIMARY OUTCOMES:
Grade of symptoms improved with early intervention. | only during RT (7WEEKS)
  using CTCAE v.5

SECONDARY OUTCOMES:
compliance on the mobile. | Only during RT (7WEEKS)
  number of reports.

CONTACTS AND LOCATIONS:
Locations (1):
- King Hussein Cancer Center, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No